CLINICAL TRIAL: NCT05638438
Title: Efficacy and Safety of the Combination of Transarterial Therapies With Donafenib Plus Anti-PD-1 Antibody for Unresectable Hepatocellular Carcinoma: A Retrospective Real-world Study
Brief Title: Efficacy and Safety of Transarterial Therapies+Donafenib + Anti-PD-1 Antibody for uHCC: A Retrospective Real-world Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-KY-180-01
Record Dates: First submitted 2022-11-27; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Hepatocellular Carcinoma Non-resectable
MeSH Terms: interventions — donafenib; spartalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: transarterial therapies — transarterial therapies combine with donafenib and Anti-PD-1 Antibody
  Other Names: donafenib; Anti-PD-1 Antibody

SUMMARY:
This Retrospective Real-world study was designed to evaluate the clinical efficacy and safety of the Combination of transarterial therapies with donafenib plus Anti-PD-1 Antibody for Unresectable Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
Data of Patients who have received Triplet therapy ( transarterial therapies+donafenib+Anti-PD-1 Antibody）will be collected，excluding incomplete data.

The primary endpoint was the objective response rate (ORR)，Secondary endpoints included disease control rate (DCR), progression-free survival rate (PFSR) [ Time Frame: 6- and 12-month], overall survival rate (OSR) [ Time Frame: 6- and 12-month], the median progression-free survival time (mPFS) and median overall survival time (mOS)， as well as adverse event.

ELIGIBILITY:
Inclusion Criteria:

1. clinically or histopathologically diagnosed HCC;
2. not suitable for curative surgery, or local ablation;
3. age 18~75 years；
4. Barcelona Clinic Liver Cancer (BCLC) Stage-B or C HCC; 5) Child-Pugh score A or B7; 6) Eastern Cooperative Group (ECOG) performance status ≤1.;

7）no serious heart, lung, or renal dysfunction； 8）at least 1 measurable lesion according to modified Response Evaluation Criteria in Solid Tumors (mRECIST)

Exclusion Criteria:

1）comorbidity with other severe systemic diseases; 2）life expectancy is less than 3 months; 3) discontinuation of treatment for personal reasons or inability to tolerate; 4）incomplete data.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Unresectable Hepatocellular Carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-02 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
the objective response rate (ORR) | From date of begining triplet therapy until disease progression or unacceptable toxicity (max 24 months)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST

SECONDARY OUTCOMES:
disease control rate (DCR) | From date of begining triplet therapy until disease progression or unacceptable toxicity (max 24 months)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST
The progression-free survival rate (PFSR) | From date of begining triplet therapy to the date of first documentation of disease progression or death, whichever occurs first (max 24 months)
  PFSR is defined as the percentage of participants who have not accured disease progression or death at the time of 6 or 12 months as assessed by RECIST 1.1 and mRECIST
The overall survival rate (OSR) | From date of begining triplet therapy to the date of first documentation of death from any cause, whichever occurs first (max 24 months)
  OSR is defined as the percentage of participants who still alive at the time of 6 or 12 months.
The progression-free survival time (mPFS) | From date of begining triplet therapy to the date of first documentation of disease progression or death, whichever occurs first(max 24 months)
  The progression-free survival time (mPFS) defined as the time from begining triplet therapy to the date of first documentation of disease progression as assessed by RECIST 1.1 and mRECIST
The median overall survival time (mOS) | From the start date of the Treatment until date of death from any cause (max 24 months)
  OS is measured from the start date of the Treatment (date of begining triplet therapy) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes earlier.
Adverse events | From the begining triplet therapy until date of death from any cause (max 24 months)
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Mingxin Pan, Prof., Principal Investigator — Southern Medical University, China